CLINICAL TRIAL: NCT03188224
Title: An App-based Transition Toolkit Targeting Youth With Chronic Health Conditions: A Randomized Trial as a Foundation to Improve Healthcare Transition and Outcomes
Brief Title: Apply the (MyTransition) App In Transition
Acronym: ApplyIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Hamilton Academic Health Sciences Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ApplyIT Study
Record Dates: First submitted 2017-06-13; First posted 2017-06-15 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Chronic Health Condition
Keywords: Transition; Improved patient outcomes; RCT; Child health; Empower youth

STUDY DESIGN:
Intervention Model Description: After completing the baseline assessment, participants will be randomized into one of two groups: intervention or control. Those in the control group will be thanked for their time and informed that the research coordinator will be in touch to set up the follow-up visits (3- and 6-months following baseline). Those in the intervention group will be provided access to the MyTransition app (intervention). The research coordinator will help them navigate through the app and will instruct them on how to use it. These participants will also receive monthly reminder messages from the research coordinator to promote the use of the app.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): MyTransition app
  Interventions: Other: MyTransition app
- Control (No Intervention): Usual care

INTERVENTIONS:
Other: MyTransition app — MyTransition app is designed to support youth moving from pediatric to adult healthcare.
  Arms: Intervention

SUMMARY:
Moving from child care to adult care is a hard time for patients and their families. Parents of children with chronic conditions say they need more support around the time of changing care. Care providers say they do not have the tools to provide smooth transitions or help their patients manage their own health. This study is to see if a smart-phone-based app (named MyTransition) can improve healthcare transition experiences and health outcomes for youth, compared to usual care.

DETAILED DESCRIPTION:
Transition to adult care is an unavoidable and challenging period for patients and their families, and comes with adverse outcomes in experience of care, population health, and costs. Parents of children with chronic conditions report a greater need for support around the time of healthcare transition. Providers report neither having the tools nor appropriate resources to foster smooth transitions for patients and their families. We hypothesize that an app-based transition toolkit (named MyTransition) designed to support youth moving from child to adult care can improve their experiences and lead to better health. The main objective of this study is to collect information to design a large multi-centre randomized control trial to assess implementation of the MyTransition app including recruitment, completion of follow-up, and scale-ability of the intervention. The secondary objective is to assess the feasibility and potential effect of the MyTransition app-based transition toolkit for improving health of youth (quality of life), healthcare transition experience, and achievement of health and life goals.

ELIGIBILITY:
Inclusion Criteria:

* Attending participating clinic at McMaster Children's Hospital
* Diagnosed with chronic health condition
* Must be able to utilize the intervention tool
* Must be able to read and understand English

Exclusion Criteria:

* Dependence on caregivers in areas of daily functioning, self-care and/or communication
* Inability to lead or provide own care
* Enrolled in a potentially confounding trial

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 39 (Actual)
Dates: Start 2018-01-25 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
Completion of Data Collection | 6-Month Follow-Up
  Completion rate of 90% for all outcomes.

SECONDARY OUTCOMES:
Change in Short Form Six-Dimension (SF-6D) | Baseline, 3-month follow-up, 6-month follow-up
  Instrument for describing and valuing individual's health. Will be used to evaluate quality of life.

OTHER OUTCOMES:
Change in Client Satisfaction Questionnaire (CSQ-8) | Baseline, 3-month follow-up, 6-month follow-up
  Designed to measure satisfaction with health and human services received by individuals and families. Will be used to assess healthcare transition experience.
Change in Transition-Q | Baseline, 3-month follow-up, 6-month follow-up
  Measures transition readiness/self-management ability. Will be used to evaluate readiness for transition.
Change in Transition Readiness Assessment Questionnaire (TRAQ) | Baseline, 3-month follow-up, 6-month follow-up
  Patient-centered questionnaire that providers and families use to assess youths' ability to make appointments, to understand their medications, and to develop other skills needed for transition to adult care. Will be used to evaluate readiness for transition.
Change in Canadian Occupational Performance Measure (COPM) | Baseline, 3-month follow-up, 6-month follow-up
  Designed to measure satisfaction with health and human services received by individuals and families. Will be used to determine achievement of health and life goals.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Willem Gorter, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster Children's Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No